CLINICAL TRIAL: NCT02360800
Title: Randomized Prospective Comparison of Tisseel Or Control to Diminish Blood Loss After Redo Redo Cardiac Surgery: the Study
Brief Title: Trial Comparing Tisseel as an Adjunct to Traditional Hemostasis After Redo Cardiac Surgery
Acronym: RETICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2015-01-14; First posted 2015-02-11 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Hemorrhage
Keywords: Bleeding; Heart Surgery; Reoperation
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TISSEEL (Experimental): Spray Fibrin Sealant
  Interventions: Procedure: Spray Fibrin Sealant
- CONTROL (Active Comparator): Traditional hemostasis and chest closure routine
  Interventions: Procedure: Traditional Hemostasis and chest Closure Routine

INTERVENTIONS:
Procedure: Spray Fibrin Sealant — Baxter Tisseel (Fibrin Sealant) is sprayed in the mediastinum at the end of the operation afetr routine chest hemostasis protocol has been completed, right before closing the chest.
  Other Names: TISSEEL
  Arms: TISSEEL
Procedure: Traditional Hemostasis and chest Closure Routine — Routine chest hemostasis and closure protocol (gauzes and inspection till satisfactory according to the surgeon)
  Arms: CONTROL

SUMMARY:
Bleeding after redo cardiac surgery is a common, unresolved and consequences-heavy event as per present day. Tisseel (Baxter inc) sprayed on the already hemostased mediastinum jut before closing seems a promising technique to radically diminish bleeding.

This study aims to verify this efficacy volume in chest drains) and possibly the consensual blood transfusion lessening.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any kind of redo cardiac surgery with ati least one previous sternotomy

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2018-09-16 (Actual)

PRIMARY OUTCOMES:
Bleeding (Amount of blood (ml) collected in chest drainage) | first 24 hours after surgery
  Amount of blood (ml) collected in chest drainage in the first 24 hours after operation

SECONDARY OUTCOMES:
Allogeneic blood Sparing (Amount of Allogeneic Blood units (number) transfused in the first 4 days after surgery) | 4 days after surgery
  Amount of Allogeneic Blood units (number) transfused in the first 4 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Lazio, Italy